CLINICAL TRIAL: NCT07092813
Title: A Phase 1, Multi-Center, Open-Label Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Sulopenem Etzadroxil + Probenecid in Adolescent Patients With Bacterial Infection
Brief Title: Pharmacokinetics of Sulopenem Etzadroxil Plus Probenecid in Adolescents
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Iterum Therapeutics, International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IT001-109
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Pharmacokinetics After Oral Intake
Keywords: Pharmacokinetics; Adolescents; Sulopenem etzadroxil; Probenecid; Sulopenem; Phase 1
MeSH Terms: interventions — Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral sulopenem (Experimental): Single dose of 500 mg of sulopenem etzadroxil and 500 mg of probenecid given orally as a bilayer tablet.
  Interventions: Drug: sulopenem etzadroxil and probenecid

INTERVENTIONS:
Drug: sulopenem etzadroxil and probenecid — single dose of 500 mg of sulopenem etzadroxil and 500 mg of probenecid given orally as a bilayer tablet.
  Other Names: Orlynvah

SUMMARY:
The goal of this clinical trial is to evaluate the use of sulopenem etzadroxil plus probenecid in adolescent patients being treated for bacterial infection. The main questions it aims to answer are:

Is sulopenem etzadroxil plus probenecid safe to use in adolescents? Is sulopenem etzadroxil plus probenecid tolerable when used in adolescents? When ingested, what does the adolescent body do to sulopenem etzadroxil plus probenecid, in terms of the movement of the drug into, through, and out of the body.

Participants will receive standard of care antibiotics for their bacterial infection as directed by their physician. In addition, participants will be asked to take a single oral dose of sulopenem etzadroxil plus probenecid. Blood samples will be collected before the dose of sulopenem etzadroxil plus probenecid, as well as at specified timepoints after the dose. Likewise, urine will be collected at specified time periods after the dose. During the course of the study, data will be collected from participants including vital sign measurements, physical examination findings, and the details of any adverse events that are reported.

DETAILED DESCRIPTION:
Sulopenem is a broad-spectrum penem β-lactam antibiotic that is being developed for the treatment of infections with common hospital and community pathogens. The intravenous (IV) formulation is intended for the initial treatment of infections in a hospital setting. ORLYNVAH (sulopenem etzadroxil and probenecid) oral tablets was approved by the FDA for the treatment of adult women with uncomplicated urinary tract infection (UTI) in October 2024. ORLYNVAH has not been studied in the pediatric population.

This is a Phase 1, multi-center, open-label study to evaluate the safety, tolerability, and pharmacokinetics (PK) of sulopenem etzadroxil plus probenecid in adolescent inpatients and outpatients that are diagnosed with bacterial infections caused by susceptible strains of Gram-positive and Gram-negative bacteria.

The primary objective of the study is to evaluate the PK of oral sulopenem etzadroxil + probenecid in adolescent inpatients and outpatients with bacterial infection. The secondary objective of the study is to evaluate the safety and tolerability of oral sulopenem etzadroxil + probenecid in adolescent inpatients and outpatients with bacterial infection.

The study will be conducted in adolescent inpatients and outpatients who are 12 to 18 years of age and are being treated for bacterial infections caused by susceptible strains (susceptible to penem antibiotics, e.g., imipenem, ertapenem, doripenem, or meropenem, and not resistant to a carbapenem) of Gram-positive and Gram-negative bacteria. Patients who meet all of the inclusion criteria and none of the exclusion criteria will be enrolled in the study. Approximately 12 patients in total will be enrolled.

On Day 1, enrolled patients will receive background antibiotic treatment other than carbapenem antibiotics, per each site's standard of care. Patients will also receive a single dose of 500 mg of sulopenem etzadroxil and 500 mg of probenecid given orally as a bilayer tablet in the fed state. This dose is the same as the approved dose for treatment of uncomplicated UTI in adult women. During treatment of the underlying bacterial infection, PK samples will be collected, and patients will be monitored for safety and tolerability. A safety follow-up will take place on Day 2 for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's parent/both parents or guardian must provide written informed consent and a statement of assent from the adolescent patient (if required by Institutional Review Board [IRB] according to local regulations and guidelines) must be obtained prior to any study-related procedures. Communication should take place between the Investigator, parent(s)/guardian, and adolescent patient to confirm understanding and compliance with the study requirements.
2. Patient is male or female adolescent who are more than or equal to 12 and <18 years of age.
3. Patient has a diagnosis of a bacterial infection as documented by the treating physician
4. Patient will be receiving appropriate anti-infective treatment for a bacterial infection.
5. Patient must have sufficient venous access to permit collection of PK samples and monitoring of laboratory safety variables.
6. Female patients who are postmenarchal must not be pregnant, or breast feeding and must have a documented negative pregnancy test at Screening.
7. Postmenarchal females and post-pubertal males must agree to use a highly effective method of birth control with partners of childbearing potential throughout the duration of the study and for 1 month following the last dose of study drug.

   NOTE: A highly effective method of birth control is defined as one that results in a low failure rate (i.e., <1% per year) when used consistently and correctly. This includes sexual abstinence, implants, some intrauterine devices, or a vasectomized partner. A vasectomy or a condom used with a spermicide is a medically acceptable form of birth control for males.
8. Patient must be willing to follow all study procedures.

Exclusion Criteria:

1. Known renal insufficiency.
2. Patient is unable to tolerate oral medications.
3. Patient has presence of any of the following conditions:

   1. Endocarditis
   2. Meningitis
   3. Necrotizing fasciitis
   4. Gas gangrene
4. Patient has signs of severe sepsis including:

   1. Shock or profound hypotension that is not responsive to fluid challenge.
   2. Disseminated intravascular coagulation as evidenced by prothrombin time or partial thromboplastin time more than or equal to 2 × the upper limit of normal (ULN) or platelets <50% of the lower limit of the normal.
5. Patient has known active liver disease or hepatic dysfunction (except a confirmed diagnosis of Gilbert's disease) defined as non-transient elevations of aspartate aminotransferase or alanine aminotransferase level elevations more than or equal to 3 × the ULN or non-transient total bilirubin more than or equal to 2 × the ULN.
6. Known neutropenia (absolute neutrophil count <500 cells/mm3).
7. Patient has history of solid organ transplantation reported at any time.
8. Patient has any finding that, in the view of the Investigator, would compromise the patient's safety requirements.
9. Patient has known allergies to penicillin, carbapenems, and/or cephalosporin antibiotics, known allergy to probenecid, or severe allergic reactions to any drug in the past.
10. Patient has a history of hypersensitivity to the study drug or any of the excipients or to medicinal products with similar chemical structures.
11. Patient or parent/legal guardian has involvement in the planning and/or conduct of this study (applies to both Iterum Therapeutics staff and/or staff at the study sites).
12. Patient has participated in any other clinical study where an investigational product was ingested within 30 days or 5 half-lives of the drug (whichever is longer) prior to the current study.
13. Patient has definite or suspected personal history or family history of clinically significant adverse drug reactions.
14. Patient has history or presence of GI, hepatic, or renal disease, or other conditions known to interfere with absorption, distribution, metabolism, or excretion of drugs.
15. Patient had treatment in the previous 3 months with any drug known to have a well-defined potential for hepatotoxicity (e.g., halothane).
16. Patient weighs <30 kg.
17. Patient is pregnant or lactating.
18. Patient has received a carbapenem as their standard of care therapy to treat the diagnosed bacterial infection.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Sulopenem plasma concentration after dose | 6 hours
  Concentrations will be determined through analysis of blood samples drawn at 1, 2, 4 and 6 hours after the dose
Probenecid plasma concentration after dose | 6 hours
  Concentrations will be determined through analysis of blood samples drawn at 1, 2, 4 and 6 hours after the dose
Sulopenem urine concentration after dose | 12 hours
  Concentrations will be determined through analysis of urine samples collected 0-2, 2-4, 4-6, 6-8 and 8-12 hours after the dose
Probenecid urine concentration after dose | 12 hours
  Concentrations will be determined through analysis of urine samples collected 0-2, 2-4, 4-6, 6-8 and 8-12 hours after dose

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events | 2 days
  Safety will be assessed by monitoring adverse events, physical examination, vital signs, and clinical laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Senior Vice President and Head of Clinical Development, Study Director — Iterum Therapeutics
Locations (1):
- Medical facility, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Pertinent individual participant data sets that underlie results in a publication are to be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Approximately July 2026 - July 2027
Access Criteria: Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. Each Investigator is obligated to keep data pertaining to the study confidential. The Investigator must consult with the Sponsor before any study data are submitted for publication. The Sponsor reserves the right to deny publication rights until mutual agreement on the content, format, interpretation of data in the manuscript, and journal selected for publication are achieved